CLINICAL TRIAL: NCT06496126
Title: Clinical Comparison of Resin-hybrid Ceramic Restorations Produced Using a Computer-aided Design/Computer-aided Manufacturing (CAD/CAM) System With Fiber-reinforced Composite Restorations
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Esmanur Kokver, Principal Investigator, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA-23074
Record Dates: First submitted 2024-06-26; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Dental Caries
Keywords: CAD/CAM; Endocrown; Fiber-reinforced composite
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cerasmart 270 (GC Coop, Tokyo, Japonya) (Experimental): Composition: Bis-MEPP, UDMA, dimethacrylate, silica (20 nm), barium glass (300 nm) 71 wt% Tooth measurement and digital design are done using a camera. The design is sent to a milling device for restoration fabrication. Tooth surface is roughened with 37% orthophosphoric acid for 10 seconds, air dried, and Adhesive Primer is applied. Inner surface of the endocrown restoration is sandblasted with aluminum oxide powder, cleaned with alcohol, and coated with Adhesive Primer. CEM ONE self-adhesive resin cement is applied to the tooth surface, and the restoration is cemented.Final polymerization process lasts 10 seconds per surface to ensure bonding.Rough edges of the restoration are polished with diamond burs and discs. Excess material is removed, and occlusion and tooth areas are checked.Any cement residues in the mouth are carefully cleaned.
  Interventions: Device: Cerasmart 270 (GC Coop, Tokyo, Japonya); Device: : G-CEM ONE (GC Coop, Tokyo, Japonya)
- EverX Flow (GC Coop, Tokyo, Japonya) (Experimental): Resin: semi-IPN matrix composed of Bis-GMA, TEGDMA and PMMA. Fillers: E-glass fiber, barium borosilicate (57 vol%) After cavity preparation, 37% phosphoric acid gel will be applied to the enamel for 30 seconds, washed with water and dried slightly. G-Premio Bond adhesive agent (GC, Tokyo, Japan) is applied to the enamel and dentin surfaces with a disposable applicator for 20 seconds and waited for 10 seconds according to the manufacturer's recommendations. Then, air is squeezed with light air pressure for 5 seconds and polymerised with LED light at 1200 mW/cm2 for 10 seconds. The restoration walls are formed with composite G-ænial™ A'CHORD (GC, Tokyo, Japan). EverX Flow composite (GC, Tokyo, Japan) is applied to the cavities in 4 mm layers and polymerised with light for 10 seconds. G-ænial™ A'CHORD (GC, Tokyo, Japan) composite is applied on the top layer. It is shaped with finishing cutters and polished with polishing rubbers.
  Interventions: Device: EverX Flow (GC Coop, Tokyo, Japonya); Device: G-Premio Bond (GC Coop, Tokyo, Japonya); Device: G-ænial A'CHORD

INTERVENTIONS:
Device: Cerasmart 270 (GC Coop, Tokyo, Japonya) — Hybrid Ceramic Block
  Arms: Cerasmart 270 (GC Coop, Tokyo, Japonya)
Device: EverX Flow (GC Coop, Tokyo, Japonya) — Fiber Reinforced Composite Resin
  Arms: EverX Flow (GC Coop, Tokyo, Japonya)
Device: : G-CEM ONE (GC Coop, Tokyo, Japonya) — Universal Self Adhesive Resin Cement
  Arms: Cerasmart 270 (GC Coop, Tokyo, Japonya)
Device: G-Premio Bond (GC Coop, Tokyo, Japonya) — Universal Adhesive
  Arms: EverX Flow (GC Coop, Tokyo, Japonya)
Device: G-ænial A'CHORD — Conventional Composite Resin
  Arms: EverX Flow (GC Coop, Tokyo, Japonya)

SUMMARY:
The aim of this clinical study was to compare the clinical performance of CAD/CAM endochrone and fibre-reinforced composite restorations in root canal treated teeth with excessive loss.

DETAILED DESCRIPTION:
Restoration of endodontically treated teeth is one of the significant challenges encountered in dentistry. The restoration of these teeth is often confronted with a series of complex factors. Following endodontic treatment, the coronal structure of the tooth may have been significantly weakened or lost. This condition makes it difficult to properly place restorative materials and restore the tooth's durability. Additionally, the weakness or loss of coronal structure after root canal treatment makes it difficult for these teeth to perform their normal functions and withstand chewing forces. Consequently, the restoration of endodontically treated teeth is a process that requires careful planning by dentists, selection of appropriate materials, and implementation of suitable techniques.

Endocrown restorations and fiber-reinforced composites (e.g., EverX Flow) are commonly used options in the restoration of such teeth. Endocrown restorations help support the tooth by covering a significant portion of the coronal structure.

GC Cerasmart 270 (GC Corporation, Tokyo, Japan) is a resin nanoceramic structure containing approximately 71% (by weight) of nanoceramic particles bonded to a resin matrix. Restorations designed digitally can be milled from a milling device for use in the production of restorations. With its enhanced strength and wear resistance, smooth restorations can be produced, limiting both aesthetic appearance and wear of opposing teeth.

Fiber-reinforced composites contain glass fibers to increase durability, thereby reducing the fragility of teeth after root canal treatment and aiding in preventing cracks. EverX Flow is a flowable composite reinforced with short fibers indicated for dentin replacement (along with a traditional composite as the enamel layer) in direct restorations and core build-ups. Due to its short fibers, EverX Flow efficiently strengthens restorations and demonstrates high fracture resistance.

In each patient, one or more endodontically treated teeth will be randomly assigned to be restored using either GC Cerasmart 270 blocks or EverX Flow (combined with GC Achord). GC Cem One Resin Cement will be used for adhesive procedures in the endocrown group, while GC G-Premio Bond will be used in the fiber composite group. Restoration procedures will be performed by a single operator. Restorations will be evaluated by two calibrated evaluators according to modified USPHS criteria at baseline and at 6 and 12 months. Data will be statistically analyzed using chi-square Cochrane and McNemar tests (p <0.05).

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals without any systemic disease
* Those between the ages of 18-65
* Individuals who brush their teeth twice a day
* Patients with at least 1 root canal treatment, loss of one or more tubercles and loss of at least 1 tooth wall in their posterior teeth after intraoral examination
* Tooth margins at gingival or supramarginal level
* Patients whose periodontal and endodontic treatments have been successfully completed and who do not show any subjective symptoms
* Voluntary individuals who agree to participate in the study and sign the informed consent form will be included in the study.
* Patients will be informed about the study, read the informed consent form and agree to be included in the study.
* Ability to apply rubber cover

Exclusion Criteria:

* Individuals with uncontrolled systemic diseases
* Individuals with mental retardation who cannot co-operate
* Individuals with advanced periodontal disease
* Individuals using removable partial dentures
* Toothache, inadequate endodontic treatment or signs of periapical lesions on clinical examination or radiographic examination
* Vital teeth
* Individuals with bruxism
* Individuals with malocclusion
* Teeth with severe loss of material that requires extraction of the relevant tooth
* Patients read the informed consent form following the information about the study and did not agree to be included in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2025-04-12 (Estimated)

PRIMARY OUTCOMES:
Retention | [Time Frame: From baseline to 24 month]
  Observers evaluated the restorations was performed using the United State Public Health Service criteria regarding retention rate. Retention rate was evaluated by 2 independent clinicians. Scores: Alfa: No loss of restorations materyal.
  Charlie: Any loss of restorative material
Marginal discoloration | [Time Frame: From baseline to 24 month]
  Observers evaluated the restorations was performed using the modified United State Public Health Service criteria regarding Marginal staining. Marginal staining was evaluated by 2 independent clinicians. Visual inspection with a mirror was performed. Scorsese: Alfa: No discoloration. Bravo: Discoloration without. Charlie:Discoloration with penetration in pulpal direction
Marginal Adaptation | [Time Frame: From baseline to 24 month]
  Observers evaluated the restorations was performed using the modified United State Public Health Service criteria regarding marginal adaptation. Marginal adaptation was evaluated by 2 independent clinicians. Visual inspection with a mirror was performed. Scores; Alfa: Closely adapted, no visible crevice. Bravo: Visible crevice, explorer will penetrate.
  Charlie: Crevice in which dentin is exposed
Seconder Caries | [Time Frame: From baseline to 24 month]
  Observers evaluated the restorations was performed using the United State Public Health Service criteria regarding retention rate. Retention rate was evaluated by 2 independent clinicians. Scores: Alfa: No caries presented. Charlie Caries present

CONTACTS AND LOCATIONS:
Overall Officials: Şükran Bolay Prof., Principal Investigator — Hacettepe University; Esmanur Kökver, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bijelic-Donova J, Myyrylainen T, Karsila V, Vallittu PK, Tanner J. Direct Short-Fiber Reinforced Composite Resin Restorations and Glass-Ceramic Endocrowns in Endodontically Treated Molars: A 4 -Year Clinical Study. Eur J Prosthodont Restor Dent. 2022 Nov 30;30(4):284-295. doi: 10.1922/EJPRD_2333Bijelic-Donova12. PMID 35438265
- [Result] Soares LM, Razaghy M, Magne P. Optimization of large MOD restorations: Composite resin inlays vs. short fiber-reinforced direct restorations. Dent Mater. 2018 Apr;34(4):587-597. doi: 10.1016/j.dental.2018.01.004. Epub 2018 Jan 20. PMID 29366492
- See also: Related info — http://www.gc.dental/europe/en-LB/products/cerasmart270
- See also: Related info — http://www.gc.dental/europe/en-LB/products/everxflow